CLINICAL TRIAL: NCT01684488
Title: A Feasibility Trial of the Youth Readiness Intervention: A Group Psychosocial Intervention for War-affected Youth in Sierra Leone
Brief Title: Trial of the Youth Readiness Intervention
Acronym: YRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: Caritas Freetown (Other); International Rescue Committee (Other); Harvard Medical School (HMS and HSDM) (Other); Yale University (Other); The City College of New York (Other)
Responsible Party: Principal Investigator, Theresa Betancourt, Salem Professor in Global Practice, Boston College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RPCGA-YRI-21003; USIP-008-10F (Other Grant/Funding Number: United States Institute for Peace)
Record Dates: First submitted 2012-03-19; First posted 2012-09-13 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Anxiety Disorder/Anxiety State; Depressive Disorder/Psychology; Social Problems/Psychology; Stress, Psychological; Violence, Non-accidental
Keywords: Depression/therapy;; Developing Countries;; Interpersonal Relations;; Life Change Events;; Psychotherapy, Group;; Resilience, Psychological;; Sierra Leone;; Survivors/psychology;; Social Adjustment;; Social Behavior;; War
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Stress, Psychological; Depression; Social Adjustment; Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Waitlist+EducAid (Active Comparator): Immediately following enrollment, participants do not immediately receive any intervention. At 3 months, they are enrolled in EducAid educational programming for the 2012-2013 academic year.
  Interventions: Other: EducAid educational programming
- Waitlist (No Intervention): Participants do not receive any intervention throughout the trial period. Once the trial has concluded, participants are invited to enroll in EducAid educational programming for the 2013-2014 academic year.
- YRI only (Experimental): Immediately following enrollment, participants complete the YRI. They are then placed on a waitlist for the remainder of the trial. At the end of the trial, participants are invited to enroll in EducAid educational programming for the 2013-2014 academic year.
  Interventions: Behavioral: YRI; Other: EducAid educational programming
- YRI+EducAid (Experimental): Immediately following enrollment, participants complete the YRI. Participants are then immediately enrolled in EducAid educational programming for the 2012-2013 academic year.
  Interventions: Behavioral: YRI; Other: EducAid educational programming

INTERVENTIONS:
Behavioral: YRI — The YRI brings together six empirically-supported practice elements shown to be efficacious across different mental health interventions, as well as methods intended to socialize youth and improve self-efficacy. Practice elements address the broad scope of problems evidenced in Sierra Leonean war-affected youth and enhance the YRI's pacing, which progresses through three phases traditionally used in trauma treatments (stabilization, integration, connection). The weekly intervention takes place over 10 sessions lasting approximately one hour and a half. Groups are divided by gender and age. Each group is paired with two interventionists of the same gender.
  Other Names: Youth Readiness Intervention
  Arms: YRI only; YRI+EducAid
Other: EducAid educational programming — EducAid is a charitable trust that provides free year-round education to over 1,500 youth, along with food, medicine, and shelter when needed. EducAid's education model aims to improve academic knowledge, self-efficacy, and attitudes toward school. Additionally, it aims to nurture hope for the future and a sense of normalcy through interactions with teachers, mentors, and peers.
  Arms: Waitlist+EducAid; YRI only; YRI+EducAid

SUMMARY:
The research will first examine data obtained from YRI participants to investigate effects of the group sessions on psychosocial and functioning outcomes in youth.

In pursuit of this aim, this research will investigate the following hypothesis: Participation in the Youth Readiness Intervention will reduce symptoms of internalizing, externalizing, trauma-related symptoms, and improve prosocial skills and functioning among war-affected 15-24 year olds in Sierra Leone.

The research also intends to examine whether youth enrolled in a psychosocial "Youth Readiness Intervention" (YRI) and a complementary education program fare better than an education-only control group, a psychosocial-only control group, and a waitlist control group.

In pursuit of this second aim, this research will investigate the following hypothesis: A combined psychosocial-education program is an effective paradigm for improving psychosocial, functional, educational, and economic self-sufficiency outcomes among war-affected youth.

DETAILED DESCRIPTION:
In Sierra Leone, a dangerous gap remains between long-term psychosocial needs and adequate services. As youth affected by the war begin to enter adulthood, they face new challenges including unemployment, interrupted education, the need to support families, marginalization and stigma, as well as the remaining psychological effects of exposure to war. Healthy social integration is critical to the long-term wellbeing of this generation, but the evidence base on effective interventions to improve skills and self-efficacy is severely limited. Despite the high burden of mental health problems among war-affected youth in Sub-Saharan Africa, few empirically-supported behavioral treatments (ESBTs) or evidence-based interventions have been implemented in this region. This study stands to make an important contribution to knowledge on effective and culturally-sensitive mental health services that can be implemented in settings fraught by multiple hardships, including war, poverty, low educational attainment, and other hardships.

This randomized study of 416 school-intending youth age 15-24 will use a parallel design to examine the potential benefits of enrolling in a psychosocial intervention--the YRI--prior to enrolling in an educational program. Assessments will be performed pre-/post-intervention and at 6-month and 12-month follow-ups. These long-term evaluations will examine whether benefits are sustained, accrue, or depreciate over time. Data will improve understanding of how a psychosocial-education intervention translates to economic outcomes like employment, as compared to an education-only intervention.

The YRI is an evidence-based group intervention developed in 2010 to address key emotional, behavioral, and functioning difficulties identified by the PI's prior longitudinal study of war-affected youth. It is designed to reduce symptoms of internalizing, externalizing, trauma-related symptoms, and improve prosocial skills and functioning among war-affected 15-24 year olds. The YRI has three overarching goals: (1) To improve interpersonal and community relationships through work with youth and community members; (2) To help vulnerable youth develop skills in emotional regulation, problem-solving, and interpersonal interactions necessary to be successful members of their communities; (3) To promote the healthy integration of difficult memories for youth who experience difficulties due to traumatic exposure. Primary mental health outcomes include decreased anxiety, hostility, and depression, and increased pro-social attitudes, as measured by the Oxford Refugee Studies Psychosocial Adjustment Scale and the African Youth Psychosocial Assessment.

EducAid is a charitable trust established in 1994. Devoted to promoting education among underprivileged and war-affected young people in Sierra Leone through holistic and academic learning, EducAid provides free year-round education to over 1,500 youth, along with food, medicine, and shelter when needed. EducAid has a keen interest in exploring how psychosocial interventions can promote academic, social, and emotional well-being in students. EducAid's education model aims to improve academic knowledge, self-efficacy, and attitudes toward school. Additionally, it aims to nurture hope for the future and a sense of normalcy through interactions with teachers, mentors, and peers. Following participation in the education component, participants' employment and economic activity will be assessed using standardized instruments for cross-cultural work, including the World Bank Living Standards Surveys.

ELIGIBILITY:
Once youth are referred to the study, a screening tool will be administered to determine whether or not they meet eligibility requirements as described below.

The screening tool contains four sections;

1. Consent and Age: assures that participants meet the age requirements
2. Oxford Refugees Psychosocial Adjustment Scale: assesses depression, anxiety and hostility
3. Functioning: assesses the participant's ability to carry out activities of daily living
4. Psychological Analysis: clinician's assessment of the psychological state of the participant.

Inclusion Criteria:

* Participants must be between 15-24 years of age;
* Participants must prefer to have the opportunity to join an educational program but not currently be enrolled in school;
* A participant's total score on the Oxford scale must equal or exceed 30 AND
* Participants must display at least one non-zero score on the functioning questions.

Exclusion Criteria:

* Participant does not plan to reside in the Freetown urban area for the duration of the study (9 months from start date);
* Participant fails to meet age requirements;
* Participant is currently enrolled in school;
* Participant is not in favor of joining an educational program;
* Participant fails to meet Oxford psychosocial or functioning thresholds;
* Participant is judged by clinical staff as:

  * Needing mental health treatment beyond the scope of the YRI
  * Otherwise not suitable for a group treatment setting
* Participant displays the following:

  * Cognitive delays
  * Active suicidality
  * Psychosis
  * Risk of harm to themselves or others

Participants at risk of harm to themselves or others, as well as those requiring treatment beyond the scope of the YRI, will be referred to local mental health or social work treatment facilities as appropriate.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 443 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in scores on the Oxford Measure of Psychosocial Adjustment & World Health Organization Disability Assessment Schedule, 2.0 (WHODAS 2.0) | Administered at 4 timepoints: (1) baseline; (2) within 15 days of YRI completion; (3) 6 months post-YRI; (4) 12 months post-YRI
  Primary outcomes of interest include changes in depression, anxiety, hostility, confidence, and pro-social behaviors. These constructs will be measured by the Oxford Refugee Studies Psychosocial Adjustment Scale. An additional primary outcome, daily functioning, will be assessed by the World Health Organization Disability Assessment Schedule, 2.0 (WHODAS 2.0). Both measures are incorporated within the study's comprehensive Youth Assessment Battery.

SECONDARY OUTCOMES:
Change in scores on the Youth Assessment Battery | Administered at 4 timepoints: (1) baseline; (2) within 15 days of YRI completion; (3) 6 months post-YRI; (4) 12 months post-YRI
  Secondary outcomes include the participant's interpersonal and community relations, experience of daily hardships, coping skills, post-traumatic stress, emotion regulation, health, risk behaviors, and other constructs as they relate to the YRI intervention areas.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa S Betancourt, ScD, MA, Principal Investigator — Boston College
Locations (1):
- CARITAS Freetown, Freetown, Sierra Leone

REFERENCES:
- [Background] Betancourt TS, Borisova II, de la Soudiere M, Williamson J. Sierra Leone's child soldiers: war exposures and mental health problems by gender. J Adolesc Health. 2011 Jul;49(1):21-8. doi: 10.1016/j.jadohealth.2010.09.021. Epub 2010 Dec 24. PMID 21700152
- [Background] Betancourt TS. Attending to the mental health of war-affected children: the need for longitudinal and developmental research perspectives. J Am Acad Child Adolesc Psychiatry. 2011 Apr;50(4):323-5. doi: 10.1016/j.jaac.2011.01.008. No abstract available. PMID 21421171
- [Background] Betancourt TS, Borisova II, Williams TP, Brennan RT, Whitfield TH, de la Soudiere M, Williamson J, Gilman SE. Sierra Leone's former child soldiers: a follow-up study of psychosocial adjustment and community reintegration. Child Dev. 2010 Jul-Aug;81(4):1077-95. doi: 10.1111/j.1467-8624.2010.01455.x. PMID 20636683
- [Background] Betancourt TS, Brennan RT, Rubin-Smith J, Fitzmaurice GM, Gilman SE. Sierra Leone's former child soldiers: a longitudinal study of risk, protective factors, and mental health. J Am Acad Child Adolesc Psychiatry. 2010 Jun;49(6):606-15. doi: 10.1016/j.jaac.2010.03.008. Epub 2010 May 1. PMID 20494270
- [Background] Betancourt TS, Agnew-Blais J, Gilman SE, Williams DR, Ellis BH. Past horrors, present struggles: the role of stigma in the association between war experiences and psychosocial adjustment among former child soldiers in Sierra Leone. Soc Sci Med. 2010 Jan;70(1):17-26. doi: 10.1016/j.socscimed.2009.09.038. Epub 2009 Oct 28. PMID 19875215
- [Background] Betancourt TS, Simmons S, Borisova I, Brewer SE, Iweala U, Soudiere MD. High Hopes, Grim Reality: Reintegration and the Education of Former Child Soldiers in Sierra Leone. Comp Educ Rev. 2008 Nov 1;52(4):565-587. doi: 10.1086/591298. No abstract available. PMID 19337570
- [Background] Betancourt TS, Bass J, Borisova I, Neugebauer R, Speelman L, Onyango G, Bolton P. Assessing local instrument reliability and validity: a field-based example from northern Uganda. Soc Psychiatry Psychiatr Epidemiol. 2009 Aug;44(8):685-92. doi: 10.1007/s00127-008-0475-1. Epub 2009 Jan 22. PMID 19165403
- [Background] Verdeli H, Clougherty K, Onyango G, Lewandowski E, Speelman L, Betancourt TS, Neugebauer R, Stein TR, Bolton P. Group Interpersonal Psychotherapy for depressed youth in IDP camps in Northern Uganda: adaptation and training. Child Adolesc Psychiatr Clin N Am. 2008 Jul;17(3):605-24, ix. doi: 10.1016/j.chc.2008.03.002. PMID 18558315
- [Background] Bolton P, Bass J, Betancourt T, Speelman L, Onyango G, Clougherty KF, Neugebauer R, Murray L, Verdeli H. Interventions for depression symptoms among adolescent survivors of war and displacement in northern Uganda: a randomized controlled trial. JAMA. 2007 Aug 1;298(5):519-27. doi: 10.1001/jama.298.5.519. PMID 17666672
- [Background] Betancourt TS, Speelman L, Onyango G, Bolton P. A qualitative study of mental health problems among children displaced by war in northern Uganda. Transcult Psychiatry. 2009 Jun;46(2):238-56. doi: 10.1177/1363461509105815. PMID 19541749
- [Background] Betancourt TS, Khan KT. The mental health of children affected by armed conflict: protective processes and pathways to resilience. Int Rev Psychiatry. 2008 Jun;20(3):317-28. doi: 10.1080/09540260802090363. PMID 18569183
- [Background] Betancourt TS. Child soldiers: reintegration, pathways to recovery, and reflections from the field. J Dev Behav Pediatr. 2008 Apr;29(2):138-41. doi: 10.1097/DBP.0b013e31816be946. No abstract available. PMID 18408537
- [Background] Betancourt TS, Williams T. Building an evidence base on mental health interventions for children affected by armed conflict. Intervention (Amstelveen). 2008;6(1):39-56. doi: 10.1097/WTF.0b013e3282f761ff. PMID 19997531
- [Derived] Betancourt TS, McBain R, Newnham EA, Akinsulure-Smith AM, Brennan RT, Weisz JR, Hansen NB. A behavioral intervention for war-affected youth in Sierra Leone: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2014 Dec;53(12):1288-97. doi: 10.1016/j.jaac.2014.09.011. Epub 2014 Oct 2. PMID 25457927
- See also: Click here for more information about this study: The Research Program on Children in Global Adversity, FXB Center, Harvard School of Public Health — http://www.harvardfxbcenter.org/programs-rpcga.php